CLINICAL TRIAL: NCT06221696
Title: Preventing Weight Regain Post-Semaglutide Treatment With Active Fiber Supplement (Soloways): A Randomized, Placebo-Controlled, Double-Blind Clinical Trial
Brief Title: Preventing Weight Regain Post-Semaglutide Treatment With Active Fiber Supplement (Soloways)
Acronym: PWR-FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other); Triangel Scientific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW005
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Overweight and Obesity
Keywords: Semaglutide; Dietary Fiber; Weight Loss; Appetite Suppression
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Fiber Supplement Group (Experimental)
  Interventions: Dietary Supplement: Active Fiber Supplement Group
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo Group

INTERVENTIONS:
Dietary Supplement: Active Fiber Supplement Group — Three daily packets of active fiber supplement (each containing 1g of glucomannan, 1g of inulin, and 3g of psyllium), taken 30 minutes before each main meal. The supplement is provided by S.Lab (Soloways), LLC.
  Arms: Active Fiber Supplement Group
Other: Placebo Group — Three daily packets of placebo powder, taken 30 minutes before each main meal.
  Arms: Placebo Group

SUMMARY:
This randomized, double-blind, placebo-controlled trial titled "Preventing Weight Regain Post-Semaglutide Treatment with Active Fiber Supplement (Soloways)" evaluated the efficacy of an active fiber supplement in preventing weight regain post-Semaglutide treatment. Participants were adults aged 18-65, with a history of obesity or overweight, and had completed a Semaglutide course. The study involved 160 participants, equally divided into two groups: one receiving the active fiber supplement (glucomannan, inulin, and psyllium) and the other a placebo, both taken 30 minutes before each main meal for 180 days. Co-primary endpoints were the percentage of weight regain from baseline to day 180 and metabolic health markers (blood glucose levels, HbA1c, lipid profile, blood pressure). Secondary endpoints included changes in BMI, body composition, and appetite assessment using VAS ratings and the Control of Eating Questionnaire (CoEQ). Participants also adhered to a reduced-calorie diet and increased physical activity, with all standard assays performed in a central laboratory. The study's objective was to determine the supplement's effectiveness in enhancing satiety, improving digestive health, and thus better managing weight compared to a placebo

ELIGIBILITY:
Inclusion Criteria:

* Adults with a history of obesity or overweight and completed Semaglutide course.
* Age 18-65 years.-

Exclusion Criteria:

* Serious chronic illnesses.
* History of bulimia or anorexia.
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of weight regain from baseline | 180 days

SECONDARY OUTCOMES:
blood glucose levels change | 180 days
blood HbA1c change | 180 days
blood total cholesterol change | 180 days
blood LDL change | 180 days
blood triglycerides change | 180 days
Systolic and diastolic blood pressure change | 180 days
BMI changes | 180 days
  Monitoring the changes in Body Mass Index from the baseline
Visceral fat rating change from baseline | 180 days
fat-free mass changes | 180 days
visceral fat changes | 180 days
total body water changes | 180 days
Effect of glucomannan, inulin, and psyllium on appetite assessed using mean postprandial participant-reported visual analog score (VAS) ratings from 0 to 10 points, where 0 is appetite absence and 10 good appetite, following a standardized breakfast | 180 days

OTHER OUTCOMES:
Fasting and mean postprandial changes in visual analog score (VAS) ratings from 0 to 10 points for thirst, nausea, and well-being following a standardized breakfast. | 180 days
Participant-reported control of eating evaluated using the Control of Eating Questionnaire (CoEQ) with 20 questions containing 5 oprions where 1 means the best and 5 the worst outcome | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia